CLINICAL TRIAL: NCT05120895
Title: A Multicenter, Prospective, Non-interventional Observational Study to Investigate the Change in Blood Cholesterol With Mevalotin® Tablet Administration in Korean Menopausal Women Aged 50 Years or More Who Require Treatment of Dyslipidemia
Brief Title: An Observational Study Investigating the Change in Blood Cholesterol With Mevalotin® Tablet Administration in Korean Menopausal Women Aged 50 Years or More Who Require Treatment of Dyslipidemia
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MVT-OS-21-01
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia; Mevalotin®; Menopause; Blood cholesterol
MeSH Terms: conditions — Dyslipidemias | interventions — Pravastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mevalotin: Korean menopausal women aged 50 years or more who required treatment of dyslipidemia and received Mevalotin® tablets.
  Interventions: Drug: Mevalotin

INTERVENTIONS:
Drug: Mevalotin — Oral tablets (starting dose 5 mg)

SUMMARY:
This study will investigate the efficacy and safety based on the observation of the blood cholesterol change with Mevalotin® Tablet administration in Korean menopausal women aged 50 years or more who require treatment of dyslipidemia.

DETAILED DESCRIPTION:
In this prospective, observational study, patient data (eg, clinical outcomes in actual clinical settings, demographic information, medical treatment-related information, Mevalotin® Tablet administration start date [Index date], and the lipid profile results at Week 24 after Mevalotin® Tablet administration start date) will be collected from medical records. No study drug will be administered in this study.

Patient data will be used to determine the change in blood cholesterol with Mevalotin® Tablet administration (5 mg, 10 mg, 20 mg, 40 mg as determined by Investigator in clinical practice) in Korean menopausal women aged 50 years or more who require treatment of dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women aged 50 years or more diagnosed with dyslipidemia

  * Menopause was defined as the condition of not having menstruation for 1 year with no specific cause or being diagnosed with menopause at the discretion of an investigator (except for the case of being diagnosed with menopause for a surgical reason within 5 years), and the menopausal status is confirmed as of the Mevalotin® Tablet administration start date (Index date).
* Patients who are determined to be prescribed with Mevalotin® Tablet at the discretion of an investigator or patients who started Mevalotin® Tablet administration within 6 weeks prior to enrollment in this observational study (however, in case of patients switching from statins to Mevalotin® Tablet, only those who receive from low/intermediate intensity statins treatment to low/intermediate intensity statins treatment can be enrolled in this study)
* Patients who provided voluntary written consent to take part in this observational study

Exclusion Criteria:

* Patients with a history of cancer within 5 years (however, patients with a history of brain tumor, breast cancer, uterine cancer, ovarian cancer, or endometrial cancer are excluded from enrollment regardless of duration.)
* Patients who received hormone replacement therapy within 1 year of enrollment
* Patients who are determined to be ineligible for participation in this observational study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Korean women are eligible for this study.
Study Population: The study population will include Korean menopausal women aged 50 years or more who are prescribed with Mevalotin® Tablet at the medical discretion of an investigator as part of routine medical practice.
Sampling Method: Non-Probability Sample
Enrollment: 3060 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in low-density lipoprotein cholesterol at Week 24 after Mevalotin® Tablet administration | Week 24 post-dose
  The change from baseline (mg/dL) in low-density lipoprotein cholesterol (LDL-C) will be assessed at Week 24 from blood plasma samples.

SECONDARY OUTCOMES:
Change from baseline in total cholesterol, triglyceride, high-density lipoprotein cholesterol, and non-high-density lipoprotein cholesterol at Week 24 after Mevalotin® Tablet administration | Week 24 post-dose
  The change from baseline (mg/dL) in total cholesterol, triglyceride, high-density lipoprotein, and non-high-density lipoprotein cholesterol will be assessed at Week 24 from blood plasma samples.
Percent change from baseline in low-density lipoprotein, total cholesterol, triglyceride, high-density lipoprotein cholesterol, and non-high-density lipoprotein cholesterol at Week 24 after Mevalotin® Tablet administration | Week 24 post-dose
  The percent change from baseline (%) in low-density lipoprotein, total cholesterol, triglyceride, high-density lipoprotein, and non-high-density lipoprotein cholesterol will be assessed at Week 24 from blood plasma samples.
Change from baseline in low-density lipoprotein, total cholesterol, triglyceride, high-density lipoprotein cholesterol, and non-high-density lipoprotein cholesterol at Week 48 after Mevalotin® Tablet administration | Week 48 post-dose
  The change from baseline (mg/dL) in total cholesterol, triglyceride, high-density lipoprotein, and non-high-density lipoprotein cholesterol will be assessed at Week 48 from blood plasma samples.
Percent change from baseline in low-density lipoprotein, total cholesterol, triglyceride, high-density lipoprotein cholesterol, and non-high-density lipoprotein cholesterol at Week 48 after Mevalotin® Tablet administration | Week 48 post-dose
  The percent change from baseline (%) in low-density lipoprotein, total cholesterol, triglyceride, high-density lipoprotein, and non-high-density lipoprotein cholesterol will be assessed at Week 48 from blood plasma samples.
Number of participants with treatment-emergent adverse events after Mevalotin® Tablet administration | Week 48 post-dose
  Treatment-emergent adverse event (TEAE) is defined as an event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (58):
- South Korea (58):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Bucheon Sejong Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital - Site 0011, Busan
  - Inje University Haeundae Paik Hospital - Site 0031, Busan
  - Boneseng Memorial Hospital, Busan
  - Pusan National University Hospital - Site 0013, Busan
  - Pusan National University Hospital - Site 0033, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Hallym University Medical Center - Chuncheon, Chuncheon
  - Kangwon National University Hospital - Site 0050, Chuncheon
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Hospital, Daegu
  - Eulji University Hospital - Site 0004, Daejeon
  - Eulji University Hospital - Site 0040, Daejeon
  - Konyang University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Myongji Hospital, Goyang-si
  - Hanyang University Guri Hospital - Site 0022, Guri-si
  - Hanyang University Guri Hospital - Site 0044, Guri-si
  - Hanyang University Guri Hospital - Site 0049, Guri-si
  - Chonnam National University Hospital Hwasun Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Pohang St. Mary's Hospital, Pohang
  - SM Christianity Hospital, Pohang
  - Bundang Jesaeng Hospital, Seongnam-si
  - Seoul National University Bundang Hospital - Site 0001, Seongnam-si
  - Seoul National University Bundang Hospital - Site 0019, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - VHS Medical Center - Site 0020, Seoul
  - VHS Medical Center - Site 0039, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital - Site 0018, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital - Site 0024, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Gwangmyeong Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Hallym University Medical Center-Kangnam, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Ajou University Hospital, Suwon
  - Uijeongbu Eulji Medical Center, Eulji University - Site 0053, Uijeongbu-si
  - Uijeongbu Eulji Medical Center, Eulji University, Uijeongbu-si
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan Univeristy Hospital, Ulsan
  - Yonsei University, Wonju Severance Christian Hospital - Site 0051, Wŏnju
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan
  - Yonsei University Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: No